CLINICAL TRIAL: NCT04306887
Title: A Open-label, Single-arm Phase Ⅱ Clinical Trial of TQ-B3101 in Subjects With Relapsed/Refractory Anaplastic Large Cell Lymphoma (ALCL)
Brief Title: A Study of TQ-B3101 in Subjects With Relapsed or Refractory Anaplastic Large Cell Lymphoma (ALCL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3101-II-02
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Relapsed/Refractory Anaplastic Large Cell Lymphoma (ALCL)
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3101 (Experimental): TQ-B3101 capsule administered orally.
  Interventions: Drug: TQ-B3101 capsule

INTERVENTIONS:
Drug: TQ-B3101 capsule — Escalating doses starting at 200 mg bid.

SUMMARY:
The objective of this study is to evaluate efficacy and safety of TQ-B3101 in subjects with relapsed/refractory anaplastic large cell lymphoma (ALCL) .

ELIGIBILITY:
Inclusion Criteria:

-1.Female or male, 10 years and older. 2.Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2. 3.Histologically or cytologically confirmed ALK positive relapsed or refractory Anaplastic Large Cell Lymphoma.

4.At least one measurable lesion. 5.Life expectancy ≥ 3 months. 6.Adequate organ system function. 7.Understood and signed an informed consent form.

Exclusion Criteria:

* 1.Primary cutaneous anaplastic large cell lymphoma. 2.Other malignancies occurred within 5 years, with exception of cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors.

  3.Has received ALK inhibitor. 4.Has received an allogeneic stem cell transplant. 5.Has received autologous stem cell transplant within 12 weeks before the first administration.

  6.Has received other anti-tumor medications within 4 weeks of the first administration.

  7.Has received major surgery within 4 weeks before the first administration. 8.Has received any curative radiotherapy or minor surgery within 2 weeks before the first administration.

  9.Has received palliative radiation therapy within 2 days before the first administration.

  10.Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1.

  11.Has uncontrollable congestive heart failure. 12.According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-29 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Baseline up to 18 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) according to Lugano response criteria.

SECONDARY OUTCOMES:
Progression free survival (PFS) within 2-year | Baseline up to 24 months
  PFS was defined as the time from the date of study enrollment to the date of the first of the following events, objective disease progression or death due to any cause.
Overall survival (OS) within 2-year | Baseline up to 24 months
  OS was defined as the time from the date of study enrollment to the date of death due to any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China